CLINICAL TRIAL: NCT05140837
Title: Early Diagnosis and Timely Treatment of Cirrhotic Patients With Minimal Hepatic Encephalopathy (CHESS-NCRCID 2106)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Collaborators: The First Affiliated Hospital of Anhui Medical University (Other); Beijing Ditan Hospital (Other); Chongqing Public Health Medical Treatment Center (Unknown); Meng Chao Hepatobiliary Hospital of Fujian Medical University (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other); Shenzhen Third People's Hospital (Other); Guizhou people's Hospital (Unknown); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Xiangya Hospital of Central South University (Other); The Second Affiliated Hospital of Hainan Medical University (Other); The Third Affiliated Hospital of Hebei Medical University (Unknown); The Second Affiliated Hospital of Harbin Medical University (Other); Henan Provincial People's Hospital (Other); Ganzhou Fifth People's Hospital (Unknown); The First Hospital of Jilin University (Other); Jiangsu People's Hospital (Unknown); First Hospital of China Medical University (Other); The Second Affiliated Hospital of Baotou Medical College (Other); Ningxia Medical University General Hospital (Unknown); The Fourth People's Hospital of Qinghai Province (Other); Xi'an High-tech Hospital (Unknown); The 10th People's Hospital affiliated to Tongji University (Unknown); Qilu Hospital of Shandong University (Other); The Third People's Hospital of Taiyuan (Other); Xichang People's Hospital (Unknown); Tianjin Third Central Hospital (Other); The Third People's Hospital of Tibet Autonomous Region (Unknown); Xinjiang Autonomous Region People's Hospital (Unknown); Second People's Hospital of Yunnan Province (Other); Hangzhou Xixi hospital (Unknown); LanZhou University (Other)
Responsible Party: Principal Investigator, Xiaolong Qi, Chief, Hepatopancreatobiliary Surgery Institute of Gansu Province
Other Study IDs: CHESS2106
Record Dates: First submitted 2021-10-27; First posted 2021-12-01 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Hepatic Encephalopathy; Cirrhosis
Keywords: Minimal hepatic encephalopathy; Cirrhosis; Psychometric hepatic encephalopathy score
MeSH Terms: conditions — Hepatic Encephalopathy; Fibrosis | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cross-sectional study
  Interventions: Diagnostic Test: Psychometric hepatic encephalopathy score & Stroop test
- real-world cohort study
  Interventions: Drug: Drug therapy

INTERVENTIONS:
Diagnostic Test: Psychometric hepatic encephalopathy score & Stroop test — MHE was assessed according to neuropsychological methods. Psychometric hepatic encephalopathy score include number connection test (NCT), digit-symbol test (DST), line-tracing test (LTT) and serial dotting test (SDT). Stroop test can assess psychomotor speed and cognitive flexibility by recording the interference response time between recognizing color fields and writing color names.
  Groups: cross-sectional study
Drug: Drug therapy — Real-world cohort study. The outcomes were examined and registered, so as to evaluate the relationship between therapeutic effects and health outcomes. Psychometric hepatic encephalopathy score and quality of life scale were measured at 3, 6, 12, 18 and 24 months of follow-up.
  Groups: real-world cohort study

SUMMARY:
Hepatic encephalopathy (HE) is a common complication of cirrhosis, which seriously damages the life quality of patients. As the disease progresses, 50-80% of patients with cirrhosis develop HE. Minimal hepatic encephalopathy (MHE) is a manifestation of HE, in which the patient usually has no obvious clinical symptoms and can only be detected by neuropsychological testing. Early identification and timely treatment are the keys to improve the prognosis of HE, and the diagnosis of MHE are the priority in the process of the disease intervention. Guidelines in many countries suggest that MHE does not recommend routine treatment. However, patients with cirrhosis usually have complex clinical complications, so whether timely treatment should be taken remains to be explored. The purpose of this study is to investigate the incidence of MHE in cirrhotic patients, and to establish a real-world cohort for further study on drug therapy and efficacy evaluation.

DETAILED DESCRIPTION:
According to the 2017 Global Burden of Disease study, there are 10.6 million patients with decompensated cirrhosis and 112 million patients with compensated cirrhosis worldwide. From 1990 to 2016, the number of patients with cirrhosis and chronic liver disease in China has increased from nearly 7 million (6833 300) to nearly 12 million (11 869 600), and the prevalence of all age groups increased by 44%. Hepatic encephalopathy (HE) is a common complication of cirrhosis, which seriously damages the life quality of patients. As the disease progresses, 50-80% of patients with cirrhosis develop HE. Minimal hepatic encephalopathy (MHE) is a manifestation of HE, in which the patient usually has no obvious clinical symptoms and can only be detected by neuropsychological testing. Early identification and timely treatment are the keys to improve the prognosis of HE, and the diagnosis of MHE are the priority in the process of the disease intervention. Guidelines in many countries suggest that MHE does not recommend routine treatment. However, patients with cirrhosis usually have complex clinical complications, so whether timely treatment should be taken remains to be explored. The purpose of this study is to investigate the incidence of MHE in cirrhotic patients, and to establish a real-world cohort for further study on drug therapy and efficacy evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-65 years;
2. confirmed cirrhosis based on clinical or pathological criteria;
3. no history of grade 1-4 hepatic encephalopathy;
4. with written informed consent.

Exclusion Criteria:

1. with other neurological or mental diseases (such as Alzheimer's disease, Parkinson's disease, etc.);
2. with alcohol or drug addiction and unstable vital signs;
3. with liver cancer or other malignant tumors;
4. fail to comply with psychological tests;
5. incomplete data collection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with cirrhosis
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-12-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Psychometric hepatic encephalopathy score (PHES) | 1 year
  The PHES is a battery of neuropsychological tests used in the diagnosis of minimal hepatic encephalopathy (MHE). The sum of scores for PHES ranges between +5 and -15. Patients with cirrhosis having a PHES score of <-4 SD are considered to have MHE.
Clinical decompensation and death | 2 year
  Clinically evident decompensating events (specifically ascites, variceal hemorrhage).
EuroQol Five Dimensions Questionnaire (EQ5D) | 2 year
  EQ5D is used to evaluate the quality of life. EQ-5D consists of two main parts: Descriptive System and Visual Analogue Scale. Five dimensions are used to describe the health state: Mobility, self-care, Usual Activities, Pain/Discomfort, Anxiety/Depression. A scale ranges from 0 to 100, with 0 representing "your worst imagined health" and 100 "your best imagined health." Self-rated information from respondents can be used as a quantitative indicator of health outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Sheng Wang, MD, Study Chair — National Clinical Research Center for Infectious Diseases; Xiaolong Qi, MD, Principal Investigator — LanZhou University; Jun-Liang Fu, MD, Principal Investigator — National Clinical Research Center for Infectious Diseases
Locations (31):
- China (31):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Ditan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chongqing Public Health Medical Treatment Center, Chongqing, Chongqing Municipality
  - MengChao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Shenzhen Third People's Hospital, Shenzhen, Guangdong
  - Guangxi Zhuang Autonomous Region People's Hospital, Nanning, Guangxi
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - The Second Affiliated Hospital of Hainan Medical College, Haikou, Hainan
  - The Third Affiliated Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - Jiangsu People's Hospital, Nanjing, Jiangsu
  - Ganzhou City Fifth People's Hospital, Ganzhou, Jiangxi
  - Bethune First Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Ningxia Medical University General Hospital, Yinchuan, Ningxia
  - The Fourth People's Hospital of Qinghai Province, Xining, Qinghai
  - Xi'an Hi-tech Hospital, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The 10th People's Hospital affiliated to Tongji University, Shanghai, Shanghai Municipality
  - The Third People's Hospital of Taiyuan, Taiyuan, Shanxi
  - Xichang People's Hospital, Xichang, Sichuan
  - Tianjin Third Central Hospital, Tianjin, Tianjin Municipality
  - The Third People's Hospital of Tibet Autonomous Region, Lhasa, Tibetan
  - Xinjiang Autonomous Region People's Hospital, Ürümqi, Xinjiang
  - Second People's Hospital of Yunnan Province, Kunming, Yunnan
  - Hangzhou Xixi Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Background] GBD 2017 Cirrhosis Collaborators. The global, regional, and national burden of cirrhosis by cause in 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet Gastroenterol Hepatol. 2020 Mar;5(3):245-266. doi: 10.1016/S2468-1253(19)30349-8. Epub 2020 Jan 22. PMID 31981519
- [Background] Li M, Wang ZQ, Zhang L, Zheng H, Liu DW, Zhou MG. Burden of Cirrhosis and Other Chronic Liver Diseases Caused by Specific Etiologies in China, 1990-2016: Findings from the Global Burden of Disease Study 2016. Biomed Environ Sci. 2020 Jan 20;33(1):1-10. doi: 10.3967/bes2020.001. PMID 32029053
- [Background] Xiao J, Wang F, Wong NK, He J, Zhang R, Sun R, Xu Y, Liu Y, Li W, Koike K, He W, You H, Miao Y, Liu X, Meng M, Gao B, Wang H, Li C. Global liver disease burdens and research trends: Analysis from a Chinese perspective. J Hepatol. 2019 Jul;71(1):212-221. doi: 10.1016/j.jhep.2019.03.004. Epub 2019 Mar 12. PMID 30871980
- [Background] Zimmermann M, Reichert AS. Rapid metabolic and bioenergetic adaptations of astrocytes under hyperammonemia - a novel perspective on hepatic encephalopathy. Biol Chem. 2021 Jul 30;402(9):1103-1113. doi: 10.1515/hsz-2021-0172. Print 2021 Aug 26. PMID 34331848
- [Background] Bale A, Pai CG, Shetty S, Balaraju G, Shetty A. Prevalence of and Factors Associated With Minimal Hepatic Encephalopathy in Patients With Cirrhosis of Liver. J Clin Exp Hepatol. 2018 Jun;8(2):156-161. doi: 10.1016/j.jceh.2017.06.005. Epub 2017 Jun 20. PMID 29892178
- [Background] Sharma K, Pant S, Misra S, Dwivedi M, Misra A, Narang S, Tewari R, Bhadoria AS. Effect of rifaximin, probiotics, and l-ornithine l-aspartate on minimal hepatic encephalopathy: a randomized controlled trial. Saudi J Gastroenterol. 2014 Jul-Aug;20(4):225-32. doi: 10.4103/1319-3767.136975. PMID 25038208
- [Background] Cabrera-Pastor A, Llansola M, Montoliu C, Malaguarnera M, Balzano T, Taoro-Gonzalez L, Garcia-Garcia R, Mangas-Losada A, Izquierdo-Altarejos P, Arenas YM, Leone P, Felipo V. Peripheral inflammation induces neuroinflammation that alters neurotransmission and cognitive and motor function in hepatic encephalopathy: Underlying mechanisms and therapeutic implications. Acta Physiol (Oxf). 2019 Jun;226(2):e13270. doi: 10.1111/apha.13270. Epub 2019 Mar 22. PMID 30830722
- [Background] Wang JY, Zhang NP, Chi BR, Mi YQ, Meng LN, Liu YD, Wang JB, Jiang HX, Yang JH, Xu Y, Li X, Xu JM, Zhang G, Zhou XM, Zhuge YZ, Tian DA, Ye J, Liu YL. Prevalence of minimal hepatic encephalopathy and quality of life evaluations in hospitalized cirrhotic patients in China. World J Gastroenterol. 2013 Aug 14;19(30):4984-91. doi: 10.3748/wjg.v19.i30.4984. PMID 23946605
- [Background] Xu XY, Ding HG, Li WG, Jia JD, Wei L, Duan ZP, Liu YL, Ling-Hu EQ, Zhuang H, Hepatology CSO, Association CM. Chinese guidelines on management of hepatic encephalopathy in cirrhosis. World J Gastroenterol. 2019 Sep 28;25(36):5403-5422. doi: 10.3748/wjg.v25.i36.5403. PMID 31576089
- [Background] Flud CR, Duarte-Rojo A. Prognostic Implications of Minimal/Covert Hepatic Encephalopathy: Large-scale Validation Cohort Studies. J Clin Exp Hepatol. 2019 Jan-Feb;9(1):112-116. doi: 10.1016/j.jceh.2018.04.009. Epub 2018 May 4. PMID 30765944
- [Background] Bajaj JS, Lauridsen M, Tapper EB, Duarte-Rojo A, Rahimi RS, Tandon P, Shawcross DL, Thabut D, Dhiman RK, Romero-Gomez M, Sharma BC, Montagnese S. Important Unresolved Questions in the Management of Hepatic Encephalopathy: An ISHEN Consensus. Am J Gastroenterol. 2020 Jul;115(7):989-1002. doi: 10.14309/ajg.0000000000000603. PMID 32618647
- [Background] Reuter B, Walter K, Bissonnette J, Leise MD, Lai J, Tandon P, Kamath PS, Biggins SW, Rose CF, Wade JB, Bajaj JS. Assessment of the spectrum of hepatic encephalopathy: A multicenter study. Liver Transpl. 2018 May;24(5):587-594. doi: 10.1002/lt.25032. PMID 29457869
- [Derived] Li XY, Liu SH, Liu C, Zu HM, Guo XQ, Xiang HL, Huang Y, Yan ZL, Li YJ, Sun J, Song RX, Yan JQ, Ye Q, Liu F, Huang L, Meng FP, Zhang XN, Yang SS, Hu SJ, Ruan JG, Li YL, Wang NN, Cui HP, Wang YM, Lei C, Wang QH, Tian HL, Qu ZS, Yuan M, Shi RC, Yang XT, Jin D, Su D, Liu YJ, Chen Y, Xia YX, Li YZ, Yang QH, Li H, Zhao XL, Tian ZM, Yu HJ, Zhang XJ, Wu CX, Wu ZJ, Li SS, Shen Q, Liu XM, Hu JP, Wu MQ, Dang T, Wang J, Meng XM, Wang HY, Jiang ZY, Liu YY, Liu Y, Qu SX, Tao H, Yan DM, Liu J, Fu W, Yu J, Wang FS, Qi XL, Fu JL. [Impact of different diagnostic criteria for assessing mild micro-hepatic encephalopathy in liver cirrhosis: an analysis based on a prospective, multicenter, real-world study]. Zhonghua Gan Zang Bing Za Zhi. 2023 Sep 20;31(9):961-968. doi: 10.3760/cma.j.cn501113-20220602-00298. Chinese. PMID 37872092